CLINICAL TRIAL: NCT04828343
Title: A Randomized, Participant-Blind, Investigator-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Rozanolixizumab Administered Subcutaneously Via Manual Push Versus Syringe Driver to Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Rozanolixizumab Administered Subcutaneously Via Manual Push Versus Syringe Driver to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP0106
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy Study Participants
Keywords: Healthy Study Participants; Phase 1; rozanolixizumab; manual push; syringe driver
MeSH Terms: interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a participant-blind and investigator-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 <50 kg (Experimental): Study participants randomized to Cohort 1 will receive a single dose of rozanolixizumab (RLZ) or placebo (PBO) subcutaneously administered with a syringe driver.
  Interventions: Drug: rozanolixizumab; Other: Placebo
- Cohort 2 <50 kg (Experimental): Study participants randomized to Cohort 2 will receive a single dose of rozanolixizumab (RLZ) or placebo (PBO) subcutaneously administered by manual push.
  Interventions: Drug: rozanolixizumab; Other: Placebo
- Cohort 3 >=50 kg (Experimental): Study participants randomized to Cohort 3 will receive a single dose of rozanolixizumab (RLZ) or placebo (PBO) subcutaneously administered with a syringe driver.
  Interventions: Drug: rozanolixizumab; Other: Placebo
- Cohort 4 >=50 kg (Experimental): Study participants randomized to Cohort 4 will receive a single dose of rozanolixizumab (RLZ) or placebo (PBO) subcutaneously administered by manual push.
  Interventions: Drug: rozanolixizumab; Other: Placebo

INTERVENTIONS:
Drug: rozanolixizumab — Study participants will receive a single dose rozanolixizumab subcutaneously administered by manual push or a syringe driver.
  Other Names: RLZ
Other: Placebo — Study participants will receive a single dose placebo subcutaneously administered by manual push or a syringe driver.
  Other Names: PBO

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of a single subcutaneous (SC) dose of rozanolixizumab administered to healthy participants by manual push (MP) versus (vs) syringe driver.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be 18 to 65 years of age, inclusive
* Study participants who are overtly healthy in the opinion of the investigator as determined by medical evaluation including medical history, a general clinical examination, including physical examination and laboratory tests, and cardiac monitoring
* Study participant has blood pressure (BP) and pulse within normal range in a supine position after 5 minutes of rest (systolic BP: 90 to 140 mmHg, diastolic BP: 50 to 90 mmHg, pulse: 40 to 90 beats per minute (bpm))
* Study participant has clinical laboratory test results within the reference ranges of the testing laboratory or not clinically significant if outside the specified ranges, in the opinion of the investigator
* Study participant's electrocardiogram (ECG) is considered "normal" or "abnormal but clinically nonsignificant" (as interpreted by the investigator)
* Study participants may be male or female
* Participant has a body mass index of 18 to 32 kg/m^2, with a minimum body weight of 35 kg

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders. Has active neoplastic disease or history of neoplastic disease within the previous 5 years of entry in the clinical study (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care approaches). Has a history of a major organ transplant or hematopoietic stem cell/marrow transplant
* Symptomatic herpes zoster within 3 months prior to Screening
* Allergies to humanized monoclonal antibodies
* Female who is pregnant or lactating
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination
* Predicted inability to comply with being free of caffeine and ethanol from 72 hours prior to clinic admission and during the In-Clinic Period of the study
* Known hypersensitivity to oral paracetamol (acetaminophen)
* History of known inflammatory bowel disease, active diverticular disease, or a history of confirmed duodenal, gastric, or esophageal ulceration in the previous 6 months
* History of hyperprolinemia, since L-proline is a constituent of rozanolixizumab.
* Twelve-lead ECG with abnormalities considered to be clinically significant upon medical review
* Renal impairment, defined as a creatinine concentration in serum of ≥1.4 mg/dL (≥123 μmol/L) for female participants and ≥1.5 mg/dL (≥132 μmol/L) for male participants
* Known viral hepatitis (B and C) or human immunodeficiency virus 1/2 antibodies or has a past medical history or family history of primary immunodeficiency or antibodies to human immunodeficiency virus type 1 and/or type 2 at Screening
* Participant has a positive test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in reverse transcriptase-polymerase chain reaction on admission to the unit
* Participant has clinical signs and symptoms consistent with SARS-CoV-2 (eg, fever, dry cough, dyspnea, sore throat, fatigue) or confirmed infection by appropriate laboratory test within the previous 14 days prior to Screening or on admission
* Participant has active infection or is symptomatic with SARS-CoV-2 or is currently in quarantine (has been in contact with a SARS-CoV-2 positive individual in the last 14 days)
* Participant has had a severe course of SARS-CoV-2 (eg, requiring extracorporeal membrane oxygenation, mechanical ventilation, or hospitalization)
* Past or intended use of over-the-counter or prescription medication (including herbal medications) within 14 days prior to dosing until Day 57
* Live vaccine(s) within 8 weeks prior to Screening or plans to receive such vaccines during the study or is within a dosing cycle to receive a second dose of a coronavirus disease-19 (COVID-19) vaccine, or within 2 weeks of having received a COVID-19 vaccine
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Exposure to more than 3 new chemical entities within 12 months prior to dosing
* Has previously been assigned to treatment in a clinical study of rozanolixizumab
* Participated in another study of an investigational medicinal product (IMP) (or a medical device) within the previous 90 days or 5 half-lives prior to Day -1 (whichever is longer) or is currently participating in another study of an IMP (or a medical device)
* Immunoglobulin G <7g/L or >16g/L at the Screening Visit
* Participant is splenectomized or has had an active clinically significant infection within the last 6 weeks
* Donated or lost >500 mL of blood or blood products in the 3 months preceding the start of dosing or plans to donate blood during the clinical study
* Employee or direct relative of an employee of the contract research organization (CRO) or UCB
* History of alcohol and/or drug abuse up to 12 months before Screening
* Smoked on average >5 cigarettes/day (or equivalent) during the last 3 months and is not able to stop smoking during the In-Clinic Period
* Excessive consumption of beverages or food containing xanthine bases (including caffeinated drinks, coffee, chocolate, etc.), equating to >400 mg caffeine per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (1):
- Up0106 001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in April 2021 and concluded in April 2022.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg): Participants with body weight greater than or equal to (>=) 35 Kilograms (kg) to less than (<) 50 kg received a single dose of rozanolixizumab (RLZ) Dose 1, subcutaneously, with a syringe driver on Day 1 of the study.
- Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg): Participants with body weight >=35 kg to <50 kg received a single dose of placebo (PBO), subcutaneously, with a syringe driver on Day 1 of the study.
- Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg): Participants with body weight >=35 kg to <50 kg received a single dose of RLZ Dose 2, subcutaneously, administered by manual push (MP) on Day 1 of the study.
- Cohort 2: Manual Push- PBO (>=35 kg to <50 kg): Participants with body weight >=35 kg to <50 kg received a single dose of PBO, subcutaneously, administered by MP on Day 1 of the study.
- Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg): Participants with body weight >=50 kg received a single dose of RLZ Dose 1, subcutaneously, with a syringe driver on Day 1 of the study.
- Cohort 3: Syringe Driver- PBO (>=50 kg): Participants with body weight >=50 kg received a single dose of PBO, subcutaneously, with a syringe driver on Day 1 of the study.
- Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg): Participants with body weight >=50 kg received a single dose of RLZ Dose 1, subcutaneously, administered by MP on Day 1 of the study.
- Cohort 4: Manual Push- PBO (>=50 kg): Participants with body weight >=50 kg received a single dose of PBO, subcutaneously, administered by MP on Day 1 of the study.
Period: Overall Study
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 3: Syringe Driver- PBO (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- PBO (>=50 kg)
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Analysis Set which consisted of all randomized study participants who received investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 3: Syringe Driver- PBO (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- PBO (>=50 kg) | Total
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (15.7) | NA (NA) — Summary statistics not reported for N<3 due to small sample size and participant identification issues. | 33.2 (9.5) | NA (NA) — Summary statistics not reported for N<3 due to small sample size and participant identification issues. | 39.3 (8.1) | NA (NA) — Summary statistics not reported for N<3 due to small sample size and participant identification issues. | 45.5 (12.7) | NA (NA) — Summary statistics not reported for N<3 due to small sample size and participant identification issues. | 37.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 6 | 2 | 2 | 0 | 2 | 1 | 21
  Male | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 1 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 6 | 2 | 0 | 0 | 0 | 0 | 13
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 2 | 1 | 0 | 0 | 4 | 2 | 4 | 2 | 15
  Other or Mixed | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 5 | 2 | 6 | 2 | 4 | 2 | 5 | 2 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) with a start date/time on or after first dose of study medication until 8 weeks after dosing of study medication.
Time Frame: From start of dosing (Day 1) to End of Safety Follow-Up (up to Day 57)
Population: The Safety Analysis Set (SS) included all randomized study participants who received IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 3: Syringe Driver- PBO (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- PBO (>=50 kg)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
percentage of participants | 83.3 | 50.0 | 100 | 50.0 | 83.3 | 0 | 83.3 | 100

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of a Single Dose Rozanolixizumab
Description: Cmax was the maximum plasma concentration of a single dose rozanolixizumab. Cmax was measured in micrograms per millilitre per milligram (ug/mL/mg).
Time Frame: Sampling time points for plasma Pharmacokinetics were as follows: predose, immediately at the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours after start of infusion, and on Days 7, 10, 13, and 16
Population: The Pharmacokinetic Per Protocol Set (PK-PPS) included all study participants who received active study medication and had at least 1 observable PK measurement and had no important protocol deviation (IPDs) affecting the PK parameters. Here, number of participants analyzed included those participants who were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL/mg
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg)
Number analyzed (Participants) | 6 | 4 | 6 | 5
ug/mL/mg | 0.03352 (52.8) | 0.004066 (127.0) | 0.007293 (644.1) | 0.02752 (82.2)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of a Single Dose Rozanolixizumab
Description: tmax was the time to maximum plasma concentration of a single dose rozanolixizumab.
Time Frame: as for outcome 2
Population: The Pharmacokinetic Per Protocol Set (PK-PPS) included all study participants who received active study medication and had at least 1 observable PK measurement and had no IPDs affecting the PK parameters. Here, number of participants analyzed included those participants who were evaluable for the outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg)
Number analyzed (Participants) | 6 | 4 | 6 | 5
hours | 60.10 [36.0 to 72.4] | 48.03 [36.0 to 72.1] | 72.00 [36.0 to 96.3] | 72.00 [36.0 to 96.1]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time t (AUC0-t) of a Single Dose Rozanolixizumab
Description: AUC0-t was the area under the plasma concentration-time curve from time zero to time t of a single dose rozanolixizumab.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ug/mL/mg
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg)
Number analyzed (Participants) | 6 | 4 | 6 | 5
hours*ug/mL/mg | 2.408 (55.4) | 0.1436 (266.7) | 0.4223 (687.0) | 2.111 (80.5)

5. Secondary Outcome: Baseline-corrected Area Under the Total Immunglobulin (Ig) G-time Curve
Description: Area under the baseline-corrected total IgG response curve from time 0 to time t.
Time Frame: Sampling time points for total IgG were as follows: 24, 36, 48, 72, and 96 hours after start of infusion, and on Days 7, 10, 13, 16, 19, 22, 29, 43 and 57
Population: Pharmacodynamic Per Protocol Set (PD-PPS) was a subset of the Safety Set (SS) which included study participants who had no IPDs affecting the PD variables, as confirmed during a pre-analysis review of the data prior to database lock. Here, number of participants analyzed included those participants who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: grams*day/Litre (g*day/L)
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 3: Syringe Driver- PBO (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- PBO (>=50 kg)
Number analyzed (Participants) | 5 | 2 | 6 | 2 | 6 | 2 | 5 | 2
grams*day/Litre (g*day/L) | -190.6 (66.10) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and standard deviation (SD) were not calculated. | -101.0 (118.4) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and SD were not calculated. | -141.8 (52.99) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and SD were not calculated. | -168.8 (49.70) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and SD were not calculated.

6. Secondary Outcome: Percent Maximum Decrease in Total Plasma IgG (Rmin) of a Single Dose Rozanolixizumab or Placebo
Description: Rmin was the maximum (max) decrease in total plasma IgG of a single dose rozanolixizumab or placebo.
Time Frame: as for outcome 5
Population: Pharmacodynamic Per Protocol Set (PD-PPS) was a subset of the Safety Set (SS) which included study participants who had no IPDs affecting the PD variables, as confirmed during a pre-analysis review of the data prior to database lock.
Measure: Mean (Standard Deviation); unit: percent max decrease in total plasma IgG
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 3: Syringe Driver- PBO (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- PBO (>=50 kg)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
percent max decrease in total plasma IgG | -46.73 (14.76) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and SD were not calculated. | -42.14 (13.31) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and SD were not calculated. | -44.03 (8.711) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and SD were not calculated. | -42.90 (10.67) | NA (NA) — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, mean and SD were not calculated.

7. Secondary Outcome: Time to Minimum IgG Level (Tmin) of a Single Dose Rozanolixizumab or Placebo
Description: tmin was the time to minimum IgG level of a single dose rozanolixizumab or placebo.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 3: Syringe Driver- PBO (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- PBO (>=50 kg)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
days | 12.08 [8.98 to 42.0] | NA [6.08 to 9.16] — As pre-specified in the SAP, if n was less than (<) 3, only the minimum and maximum were reported, median could not be calculated. | 11.07 [6.11 to 15.1] | NA [4.00 to 42.1] — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, median could not be calculated. | 9.012 [5.97 to 12.1] | NA [5.96 to 15.1] — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, median could not be calculated. | 10.55 [4.00 to 15.0] | NA [2.00 to 8.95] — As pre-specified in the SAP, if n<3, only the minimum and maximum were reported, median could not be calculated.

ADVERSE EVENTS:
Time Frame: From start of dosing (Day 1) to End of Safety Follow-Up (up to Day 57)
Description: A TEAE was defined as any AE with a start date/time on or after first dose of study medication until 8 weeks after dosing of study medication (termination or Withdrawal Visit). The Safety Analysis Set (SS) consisted of all randomized study participants who received IMP.
Arm/Group | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) | Cohort 3: Syringe Driver- PBO (>=50 kg) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) | Cohort 4: Manual Push- PBO (>=50 kg)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 5/6 | 1/2 | 6/6 | 1/2 | 5/6 | 0/2 | 5/6 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Syringe Driver- RLZ Dose 1 (>=35 kg to <50 kg) (N=6) | Cohort 1: Syringe Driver- PBO (>=35 kg to <50 kg) (N=2) | Cohort 2: Manual Push- RLZ Dose 2 (>=35 kg to <50 kg) (N=6) | Cohort 2: Manual Push- PBO (>=35 kg to <50 kg) (N=2) | Cohort 3: Syringe Driver- RLZ Dose 1 (>=50 kg) (N=6) | Cohort 3: Syringe Driver- PBO (>=50 kg) (N=2) | Cohort 4: Manual Push- RLZ Dose 1 (>=50 kg) (N=6) | Cohort 4: Manual Push- PBO (>=50 kg) (N=2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT04828343/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT04828343/SAP_001.pdf